CLINICAL TRIAL: NCT05455736
Title: STereotactic sAlvage Radiotherapy for Macroscopic Prostate Bed Recurrence After prostatectomy-a Prospective Observational Study -STARR
Brief Title: STereotactic sAlvage Radiotherapy for Macroscopic Prostate Bed Recurrence After prostatectomy-a Prospective Observational Study
Acronym: STARR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: STARR
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer; Relapse
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stereotactic salvage radiotherapy for macroscopic prostate bed relapse — Stereotactic prostate salvage radiotherapy administered on prostate bed macroscopic recurrence. Different techniques will be allowed provided that treatment respects doses and fractionation indicated per-protocol (35 Gy in 5 fractions)

SUMMARY:
STereotactic sAlvage Radiotherapy for macroscopic prostate bed Recurrence after prostatectomy (STARR trial) is a prospective observational study aimed to assess outcome after Stereotactic salvage radiotherapy (SSRT) for macroscopic prostate bed recurrence after radical prostatectomy.

DETAILED DESCRIPTION:
This is a prospective observational multicenter study including patients affected by patients with macroscopic recurrence within prostate bed after RP detected with Choline or PSMA CT-PET and confirmed with pelvic MRI (except for cases in which MRI is contraindicated). Patients will be treated with SSRT on macroscopic prostate bed recurrence for a total dose of from 35 in 5 fractions. Planned size of the overall study population is 90 patients. The study will include a screening phase and a treatment phase. The screening phase allows for assessment of subject eligibility, demographics, PSA, comorbidities and current drug therapies up to 45 days prior to randomization.

The treatment phase consists of SSRT administered on prostate bed macroscopic recurrence. Different techniques will be allowed provided that treatment respects doses and fractionation indicated per-protocol (35 Gy in 5 fractions) and that dose constraints to organs at risk (OAR) reported in this document are observed. The total planned duration of the study is 40 months, consisting in 16 months enrollment period, during which patients will perform the screening and and later phase of 24 months in which patients will continue to be submitted to periodic checks every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by biochemical recurrence after radical prostatectomy for prostate cancer (defined as a PSA increase > 0.2 ng/ml)
* Presence of macroscopic recurrence in prostate bed, determined with either Choline or PSMA PET imaging and confirmed through MRI (except for cases in which MRI is contraindicated)
* Absence of distant and/or regional sites of disease outside prostate bed
* Patients free from Androgen deprivation therapy (ADT) (Adjuvant ADT after radical prostatectomy for pN+ patients is allowed if > 12 months from biochemical recurrence)

Exclusion Criteria:

* Presence of distant and/or regional sites of disease outside prostate bed
* Patient undergoing ADT or withdrawal of adjuvant ADT within12 months from biochemical recurrence
* Absence of disease detection from one of the two imaging modalities used (Choline or PSMA Pet and MRI must be positive- except for cases in which MRI is contraindicated)
* Any condition for which, in the opinion of the treating physician, SSRT would be contraindicated for the patient (i.e peristence of moderate/severe urinary distress after prostatectomy, post-surgical complications etc)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by macroscopic prostate bed relapse
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-07-11 (Estimated); Study Completion 2024-07-11 (Estimated)

PRIMARY OUTCOMES:
Biochemical relapse free survival (BRFS) | 2 year
  Primary endpoint of the study is BRFS after treatment, biochemical relapse is defined as a PSA increase above 0.2 ng/ml for patients with a PSA nadir < 0.2 ng/ml or 2 consecutive PSA increases > 25% if compared to nadir in patients with a PSA nadir > 0.2 ng/ml.

SECONDARY OUTCOMES:
Rate of patients with complete response | at 2 years after treatment
  Complete response is defined as PSA nadir <0.2 ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi Radiation Oncology Unit, Florence, Italy